CLINICAL TRIAL: NCT00315510
Title: Does Rosuvastatin Reduce Ischemia/Reperfusion Injury in Humans In-Vivo? A Randomized Double Blind Placebo Controlled Trial
Brief Title: Rosuvastatin and Ischemia Reperfusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QPhT05_131005-Rosuvastatine
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Ischemia
Keywords: Ischemia-reperfusion; Annexin A5
MeSH Terms: conditions — Ischemia | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin

SUMMARY:
Statins, including rosuvastatin, are drugs that lower plasma cholesterol and prevent atherosclerotic disease. Recent preclinical evidence suggests that statins also increase tissue tolerance to ischemia-reperfusion injury.

This is a randomized, double blind, parallel designed study comparing the effect of 1 week treatment with rosuvastatin (20 mg, once a day) with placebo on forearm ischemia-reperfusion injury in healthy male volunteers. Forearm ischemia-reperfusion injury is quantified with Tc-99m-annexin A5 scintigraphy of the hands after a standardized ischemic exercise test. For this purpose, Tc-99m-rh-annexin A5 (400 MBq; < 5 mSv) is injected intravenously upon reperfusion, followed by scintigraphy of both hands with a gamma camera at 1 and 4 hours after injection. Annexin A5 targeting is calculated as the percentage difference in activity (counts/pixel) between the thenar muscles of both hands.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (18-50 years of age)

Exclusion Criteria:

* Hypercholesterolemia
* Hypertension

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2006-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
annexin A5 targeting to ischemically exercised hand

SECONDARY OUTCOMES:
plasma lipid levels

CONTACTS AND LOCATIONS:
Overall Officials: Gerard A. Rongen, MD, PhD, Principal Investigator — Dept. of Pharmacology-Toxicology; Radboud University Medical Centre
Locations (1):
- Clinical Research Centre Nijmegen; Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Rongen GA, Oyen WJ, Ramakers BP, Riksen NP, Boerman OC, Steinmetz N, Smits P. Annexin A5 scintigraphy of forearm as a novel in vivo model of skeletal muscle preconditioning in humans. Circulation. 2005 Jan 18;111(2):173-8. doi: 10.1161/01.CIR.0000151612.02223.F2. Epub 2004 Dec 27. PMID 15623546
- [Derived] Meijer P, Oyen WJ, Dekker D, van den Broek PH, Wouters CW, Boerman OC, Scheffer GJ, Smits P, Rongen GA. Rosuvastatin increases extracellular adenosine formation in humans in vivo: a new perspective on cardiovascular protection. Arterioscler Thromb Vasc Biol. 2009 Jun;29(6):963-8. doi: 10.1161/ATVBAHA.108.179622. Epub 2009 Apr 9. PMID 19359665